CLINICAL TRIAL: NCT02739581
Title: Efficacy and Safety of Endoscopic Variceal Ligation (EVL) Versus EVL Plus Non-selective B-blockers (NSBB) For Prevention of Variceal Rebleed and Non-bleed Related Complications in Patients With Advanced Cirrhosis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funds
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-04
Record Dates: First submitted 2016-04-12; First posted 2016-04-15 (Estimated); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Advanced Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Endoscopic variceal ligation with Non-selective B-blockers (Experimental)
  Interventions: Procedure: Endoscopic Variceal Ligation; Drug: Non selective beta blocker
- Endoscopic variceal ligation with Placebo (Active Comparator)
  Interventions: Procedure: Endoscopic Variceal Ligation; Other: Placebo

INTERVENTIONS:
Procedure: Endoscopic Variceal Ligation
Drug: Non selective beta blocker
  Arms: Endoscopic variceal ligation with Non-selective B-blockers
Other: Placebo
  Arms: Endoscopic variceal ligation with Placebo

SUMMARY:
The patients will be randomized into two groups

1. Endoscopic Variceal Ligation with Non Selective Beta Blocker
2. Placebo with Endoscopic Variceal Ligation

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 80 years old.
* Clinical criteria and/or analytical, ultrasound and/or liver biopsy consistent with the diagnosis of liver cirrhosis.
* Endoscopic Diagnosis of esophageal variceal bleeding within 5 days prior to study inclusion.
* Written informed consent to participate in the study.
* Child C status, CTP >10

Exclusion Criteria:

* Pregnancy or lactation
* Serum Creatinine > 2 mg/dl
* Bleeding due to gastric varices.
* Active infection or recent infection < 2 weeks
* Presence of hepatocellular carcinoma or portal vein thrombosis
* Active alcoholism
* Pregnancy
* HIV infection
* Severe heart, respiratory or contraindications for beta blockers(severe chronic obstructive pulmonary disease, severe asthma, severe insulin-dependent diabetes mellitus, Brady arrhythmia)
* Not giving consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Recurrence of variceal bleeding | 12 months

SECONDARY OUTCOMES:
Recurrence of variceal bleeding | 24 months
Survival | 12 months
Survival | 24 months
Bleeding severity in both arms | 12 months
Bleeding severity in both arms | 24 months
Incidence or progression of Portal Hypertension complications such as ascites control in both arms. | 12 months
Incidence or progression of Portal Hypertension complications such as Spontaneous Bacterial Peritonitis in both arms. | 12 months
Incidence or progression of Portal Hypertension complications such as Hepatorenal syndrome in both arms. | 12 months
Appearance or progression of Portal Vein Thrombosis in both arms | 12 months
Number of patients receive alternative treatments transhepatic intrajugular portosystemic shunt in both arms. | 12 months
Incidence of adverse events in both groups | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr Ankur Jindal, MD, Principal Investigator — Institute of Liver and Biliary Sciences
Locations (1):
- Institute of liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided